CLINICAL TRIAL: NCT01409161
Title: Phase II Study of Treatment of Acute Promyelocytic Leukemia (APL) With ATRA, Arsenic Trioxide and Gemtuzumab Ozogamicin (GO)
Brief Title: Tretinoin and Arsenic Trioxide With or Without Gemtuzumab Ozogamicin in Treating Patients With Previously Untreated Acute Promyelocytic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0981; NCI-2011-02767 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2010-0981 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Acute Promyelocytic Leukemia With PML-RARA
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide; arsenous acid; Gemtuzumab; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tretinoin, arsenic trioxide, gemtuzumab ozogamicin) (Experimental): INDUCTION: Patients receive tretinoin PO BID, arsenic trioxide IV over 1-2 hours daily, and gemtuzumab ozogamicin IV over 2 hours once at weeks 1-4.
  CONSOLIDATION: Patients achieving CR receive arsenic trioxide IV 5 days per week during weeks 1-4, 9-12, 17-20, and 25-28 and tretinoin PO BID for 2 weeks on and 2 weeks off. Treatment repeats every 8 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Arsenic Trioxide; Drug: Gemtuzumab Ozogamicin; Other: Laboratory Biomarker Analysis; Drug: Tretinoin

INTERVENTIONS:
Drug: Arsenic Trioxide — Given IV
  Other Names: Arsenic (III) Oxide; Arsenic Sesquioxide; Arsenous Acid; Arsenous Acid Anhydride; Arsenous Oxide; Trisenox; White Arsenic
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; gemtuzumab; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Tretinoin — Given PO
  Other Names: 2,4,6,8-Nonatetraenoic acid, 3, 7-dimethyl-9-(2,6,6-trimethyl-1-cyclohexen-1-yl)-, (all-E)-; Aberel; Airol; Aknoten; all trans-Retinoic acid; All-trans Retinoic Acid; All-trans Vitamin A Acid; all-trans-Retinoic acid; all-trans-Vitamin A acid; ATRA; Avita; beta-Retinoic Acid; Cordes Vas; Dermairol; Epi-Aberel; Eudyna; Renova; Retin-A; Retin-A MICRO; Retin-A-Micro; retinoic acid; Retisol-A; Ro 5488; Stieva-A; Stieva-A Forte; Trans Retinoic Acid; Trans Vitamin A Acid; trans-Retinoic acid; Tretinoinum; Vesanoid; vitamin A acid; Vitamin A acid, all-trans-; Vitinoin

SUMMARY:
This phase II trial studies how well tretinoin and arsenic trioxide with or without gemtuzumab ozogamicin works in treating patients with previously untreated acute promyelocytic leukemia. Drugs used in chemotherapy, such as tretinoin and arsenic trioxide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotoxins, such as gemtuzumab ozogamicin, may find certain cancer cells and kill them without harming normal cells. Giving tretinoin and arsenic trioxide together with gemtuzumab ozogamicin may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess whether a combination of all-trans retinoic acid (ATRA [tretinoin]), and arsenic trioxide (ATO) can produce long-term event-free survival in patients with low-risk untreated acute promyelocytic leukemia (APL).

II. Assess whether administration of gemtuzumab ozogamicin (GO) at the diagnosis in patients with high-risk APL (white blood cell [WBC] > 10,000) and if the WBC rises to > 10,000 after start of treatment (in patients with low-risk disease) will improve complete response (CR) rate without increasing toxicity in high-risk untreated APL.

OUTLINE:

INDUCTION: Patients receive tretinoin orally (PO) twice daily (BID), arsenic trioxide intravenously (IV) over 1-2 hours daily, and gemtuzumab ozogamicin IV over 2 hours once at weeks 1-4.

CONSOLIDATION: Patients achieving CR receive arsenic trioxide IV 5 days per week during weeks 1-4, 9-12, 17-20, and 25-28 and tretinoin PO BID for 2 weeks on and 2 weeks off. Treatment repeats every 8 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of APL based on the presence of the PML-RAR-alpha fusion gene by cytogenetics, polymerase chain reaction (PCR), or POD test
* Ability to understand and the willingness to sign a written informed consent document indicating that they are aware of the investigational nature of the study
* Patients in whom therapy for APL was initiated on an emergent basis are eligible (patients may have already started treatment with ATRA, ATO, and/or one dose of idarubicin due to the urgency to start therapy early)
* Women of child-bearing potential must have a negative serum pregnancy test at screening; in addition to having a negative pregnancy test confirmed at screening, all female participants of childbearing potential must have a negative pregnancy test confirmed within 48 hours prior to dosing with the study drug
* All sexually active subjects (males and females of child-bearing potential) agree to use 2 effective methods of contraception for the duration of the study

Exclusion Criteria:

* Fridericia corrected QT (QTcF) interval on the electrocardiogram (EKG) greater than 480 milliseconds
* Patients with creatinine > 2.5 times upper limit of normal unless felt to be related the underlying leukemia by the treating physician or hemolysis or Gilbert's disease
* Patients with total bilirubin >= 2.0 times upper limit of normal unless felt to be related the underlying leukemia by the treating physician or hemolysis or Gilbert's disease
* Patients with alanine aminotransferase (ALT)/aspartate aminotransferase (AST) > 3 times upper limit of normal unless felt to be related the underlying leukemia by the treating physician or hemolysis or Gilbert's disease

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Estimated)
Dates: Start 2011-10-05 (Actual); Primary Completion 2027-12-18 (Estimated); Study Completion 2027-12-18 (Estimated)

PRIMARY OUTCOMES:
Event free survival | The time from the start of treatment to first documentation of disease relapse or death, assessed up to 2 years
  Monitored using a Bayesian time-to-event model.

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson Regional Care Center-Katy, Houston, Texas
  - MD Anderson Regional Care Center-Bay Area, Nassau Bay, Texas
  - MD Anderson Regional Care Center-Sugar Land, Sugar Land, Texas
  - MD Anderson Regional Care Center-The Woodlands, The Woodlands, Texas

REFERENCES:
- [Derived] Jen WY, Marvin-Peek J, Kantarjian HM, Alvarado Y, Borthakur G, Jabbour E, Wierda W, Kadia TM, Daver NG, DiNardo CD, Short NJ, Jain N, Ferrajoli A, Kornblau S, Yilmaz M, Ohanian M, McCue D, Burger J, Hammond D, Patel K, Issa GC, Pemmaraju N, Sasaki K, Maiti A, Abbas HA, Chien K, Takahashi K, Haddad F, Bose P, Masarova L, Montalban-Bravo G, Swaminathan M, Brandt M, Pierce S, Garcia-Manero G, Ravandi F. Long-term follow-up of a phase 2 study of all-trans retinoic acid, arsenic trioxide, and gemtuzumab ozogamicin in acute promyelocytic leukemia. Cancer. 2025 Jan 1;131(1):e35662. doi: 10.1002/cncr.35662. Epub 2024 Nov 25. PMID 39584789
- See also: M D Anderson Cancer Center — http://www.mdanderson.org